CLINICAL TRIAL: NCT05658705
Title: Preoperative Supine Time for Adrenal Venous Sampling: A Prospective Randomized Controlled Trial
Brief Title: Preoperative Supine Time for Adrenal Venous Sampling
Acronym: PSTAVS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHZhejiangU-004
Record Dates: First submitted 2022-11-28; First posted 2022-12-21 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Primary Aldosteronism
Keywords: adrenal venous sampling; preoperative supine time; primary aldosteronism; resistant hypertension
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients and investigators cannot be blinded due to the type of study. To minimize the potential influence of this limitation, we will assign the most professional vascular doctor to perform the same operation on the two groups of patients, and statisticians will be blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group(15-min supine group) (Experimental): Participants in the experimental group will keep supine position for 15 minutes before AVS.
  Interventions: Procedure: 15-min supine time
- control group(2-hour supine group) (Active Comparator): Participants in the control group will keep supine position for 2 hours before AVS.
  Interventions: Procedure: 2-hour supine time

INTERVENTIONS:
Procedure: 15-min supine time — The length of preoperative supine time before AVS was 15 minutes.
  Arms: experimental group(15-min supine group)
Procedure: 2-hour supine time — The length of preoperative supine time before AVS was 2 hours.
  Arms: control group(2-hour supine group)

SUMMARY:
This study aim to understand whether the length of preoperative supine time would affect the AVS outcome.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is the most common form of secondary hypertension, accounting for 5% of hypertensive patients and 17-23% in patients with resistant hypertension. Compared to the primary hypertension, PA is more prone to cause severe organ damage and even early death. Adrenal venous sampling (AVS) is an effective confirmatory test for subtyping unilateral and bilateral adrenal hyperplasia, helping doctors to make an accurate decision between surgery or medication. Supine in bed before AVS is recommended for a desirable result of AVS according to guidelines. However, investigating study about the most optimal preoperative supine time before AVS is lacking. This is a single-center prospective randomized controlled study. 120 patients diagnosed as PA and with willing for further AVS examination will be included. Participants will be randomly allocated to 15-min supine time group or 2-hours supine time group. The primary outcomes are the degrees of clinical and laboratory remission (blood pressure, type and dose of antihypertensive drugs, serum potassium, orthostatic ARR). The secondary outcomes are the technical success rate and adverse event of AVS (selective index≥2 is considered as successful surgery without corticotropin stimulate). Discussion: Primary aldosteronism is an intractable public health problem, and many techniques including AVS have been developed to correctly identify this disease. This study will help to understand whether the length of preoperative supine time would affect the diagnostic efficacy of AVS, and thus help to formulate a more reasonable AVS procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are clinically diagnosed as primary aldosteronism with ARR≥37 (PAC showed as pg/ml, renin showed as μIU/mL) and passed through PA confirmatory tests (PAC-post CCT>110pg/ml, PAC-post SSIT >80pg/ml, or PAC-post FST>60pg/ml). PAC: plasma aldosterone concentration;
2. Patients with willing for AVS;
3. Age 18 or above, male or female, with legal capacity.

Exclusion Criteria:

1. Patients with suspected adrenocortical carcinoma or pheochromocytoma;
2. Patients with high risk of adrenal surgery;
3. Patients have been subtyping to glucocorticoid-suppressible hyperaldosteronism or familial hyperaldosteronism type III;
4. Patients were diagnosed as Cushing syndrome or subclinical Cushing syndrome;
5. Patients were treated with glucocorticoids recently;
6. Patients with whole body or venipuncture area infection;
7. Patients with venous access thrombosis;
8. Patients are allergic to iodine;
9. Patients with X-ray contraindications;
10. Patients with coagulation dysfunction;
11. Patients are unable to cooperate and follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-03-29 (Estimated); Study Completion 2025-03-29 (Estimated)

PRIMARY OUTCOMES:
The rate of complete biochemical remission | At 6 months of follow-up
  Compare the rate of complete biochemical remission between two groups. Blood was drawn to measure aldosterone, renin and potassium. According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes. The proportion of complete biochemical remission according to PASO consensus criteria.

SECONDARY OUTCOMES:
The rate of complete clinical remission | At 6 months of follow-up
  Compare the rate of complete clinical remission between two groups. The proportion of complete clinical remission according to PASO consensus criteria. Clinical outcomes were determined by the blood pressure response to treatment and the number and dosage of antihypertensive medications.
Successful catheterization rate | At baseline
  Intraoperative bilateral SI value was used to judge whether the blood collection cannula was successful. In the surgery absence of osyntropin, SI≥2 was used as the standard for successful blood collection and LI≥2 was used for judging the dominant side aldosterone secretion.
Adverse events | At 3 months of follow-up
  Record the occurrence of adverse events, including adrenal venous hemorrhage and related adrenal insufficiency, hypertensive urgencies, anaphylactic shock, venous thrombosis, pulmonary embolism, ect.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Zhen jie, MD,PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The second affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Background] Zhong S, Zhang T, He M, Yu H, Liu Z, Li Z, Song X, Xu X. Recent Advances in the Clinical Application of Adrenal Vein Sampling. Front Endocrinol (Lausanne). 2022 Feb 9;13:797021. doi: 10.3389/fendo.2022.797021. eCollection 2022. PMID 35222268
- [Background] Liu Z, He M, Song X, Xu F, Zhang B, Chen B, Yu P, Zhou H, Shan L, Wang H, Gu Z, Zhong S, Xu X, Tao Z, Chen B, Gu W. Computed tomography image fusion, Coaxial guidewire technique, Fast intraprocedural cortisol testing technique improves success rate and decreases radiation exposure, procedure time, and contrast use for adrenal vein sampling. J Hypertens. 2021 Sep 1;39(9):1918-1925. doi: 10.1097/HJH.0000000000002852. PMID 34039913
- [Background] Zennaro MC, Boulkroun S, Fernandes-Rosa FL. Pathogenesis and treatment of primary aldosteronism. Nat Rev Endocrinol. 2020 Oct;16(10):578-589. doi: 10.1038/s41574-020-0382-4. Epub 2020 Jul 28. PMID 32724183
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Rossi GP, Auchus RJ, Brown M, Lenders JW, Naruse M, Plouin PF, Satoh F, Young WF Jr. An expert consensus statement on use of adrenal vein sampling for the subtyping of primary aldosteronism. Hypertension. 2014 Jan;63(1):151-60. doi: 10.1161/HYPERTENSIONAHA.113.02097. Epub 2013 Nov 11. PMID 24218436
- [Background] Seccia TM, Miotto D, Battistel M, Motta R, Barisa M, Maniero C, Pessina AC, Rossi GP. A stress reaction affects assessment of selectivity of adrenal venous sampling and of lateralization of aldosterone excess in primary aldosteronism. Eur J Endocrinol. 2012 May;166(5):869-75. doi: 10.1530/EJE-11-0972. Epub 2012 Feb 13. PMID 22330150
- [Derived] He M, Zhang Y, Song X, Zhang T, Yu H, Ji Y, Gong S, Chai P, Chen J, Wang S, Chen B, Xu X, Liu Z. Preoperative supine time for adrenal venous sampling: a prospective randomized controlled trial. Trials. 2024 Jan 2;25(1):14. doi: 10.1186/s13063-023-07872-2. PMID 38167540